CLINICAL TRIAL: NCT03298399
Title: A Phase I Study of Mesenchymal Stromal Cells to Promote Stem Cell Engraftment in Patients With Severe Sickle Cell Disease Undergoing Haploidentical Hematopoietic Cell Transplantation
Brief Title: Mesenchymal Stromal Cells for Haplo Hematopoietic Cell Transplantation for Sickle Cell Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped due to a competing trial.
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elizabeth Stenger, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00090514; 1K23HL133446 (NIH)
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Sickle Cell Disease
Keywords: Hematopoietic cell transplantation (HCT); Haploidentical; Mesenchymal stromal cells
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MSC dose level 1 (Experimental): The first three subjects (minimum) will receive four weekly infusions of MSCs.
  Interventions: Biological: Autologous MSCs
- MSC dose level 2 (Experimental): If no significant side effects are encountered at dose level 1, then subsequent subjects will receive four infusions of MSCs given twice weekly.
  Interventions: Biological: Autologous MSCs
- MSC dose level 3 (Experimental): If dose level 2 is well tolerated, then subsequent subjects will receive six infusions MSCs given twice weekly.
  Interventions: Biological: Autologous MSCs

INTERVENTIONS:
Biological: Autologous MSCs — Participants at dose level 1 receive four infusions of MSCs, given once per week. The first MSC infusion will be given no sooner than 4 hours after the bone marrow transplant. The total number of cells delivered to each patient will depend on their weight and assigned dose level. The maximal individual dose of MSCs any patient will receive is 2 x 10^6 cells/kg, which will be delivered via intravenous infusion. The infusion can be administered to patients in the inpatient or outpatient setting.
  Arms: MSC dose level 1
Biological: Autologous MSCs — Participants at dose level 2 receive four infusions of MSCs, given twice per week. The first MSC infusion will be given no sooner than 4 hours after the bone marrow transplant. The total number of cells delivered to each patient will depend on their weight and assigned dose level. The maximal individual dose of MSCs any patient will receive is 2 x 10^6 cells/kg, which will be delivered via intravenous infusion. The infusion can be administered to patients in the inpatient or outpatient setting.
  Arms: MSC dose level 2
Biological: Autologous MSCs — Participants at dose level 3 receive six infusions of MSCs, given twice per week. The first MSC infusion will be given no sooner than 4 hours after the bone marrow transplant. The total number of cells delivered to each patient will depend on their weight and assigned dose level. The maximal individual dose of MSCs any patient will receive is 2 x 10^6 cells/kg, which will be delivered via intravenous infusion. The infusion can be administered to patients in the inpatient or outpatient setting.
  Arms: MSC dose level 3

SUMMARY:
This trial is being conducted as a step toward testing the long-term hypothesis that freshly cultured, autologous mesenchymal stromal cells (MSCs) grown in platelet lysate-containing medium will modulate recipient T-cell immune responses and promote engraftment in haploidentical hematopoietic cell transplant (HCT) recipients. As a phase I, dose escalation trial of autologous MSCs in patients with sickle cell disease (SCD) undergoing haploidentical HCT, the main aim is to evaluate the safety of this therapy with a secondary aim to evaluate its effects on engraftment and graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
This is a single center, phase I, open label dose escalation study designed to determine the safety and tolerability of autologous, bone marrow-derived MSCs (EPIC2016-MSC003) in patients with SCD undergoing haploidentical HCT.

Study participants are assigned to one of three MSC dose levels: four infusions of MSCs given once per week, four infusions given twice per week, or six infusions given twice per week. Bone marrow (1-2 ml/kg, max 60 ml) will be collected from study participants for autologous MSC expansion a minimum of 28 days prior to first planned MSC infusion. MSCs will be expanded ex vivo in human platelet lysate to the specified dose level. All MSC infusions will be dosed at 2 x 10^6 MSCs/kg recipient weight, with first infusion given on day 0 (day of haploidentical HCT) or day +1. This phase I trial will enroll 12-18 patients with severe SCD undergoing haploidentical HCT, with subjects followed for 1 year following HCT (and MSC infusions).

Prior to MSC infusions, study participants will undergo transplant conditioning and GVHD prophylaxis as follows:

Day -100 to -10: Hydroxyurea 30 mg/kg PO Qday

Day -9: Rabbit anti-thymocyte globulin (ATG) 0.5 mg/kg IV

Day -8: Rabbit ATG 2 mg/kg IV

Day -7: Rabbit ATG 2 mg/kg IV; Thiotepa 10 mg/kg IV

Day -6: Fludarabine 30 mg/m2 IV; Cyclophosphamide 14.5 mg/kg IV

Day -5: Fludarabine 30 mg/m2 IV; Cyclophosphamide 14.5 mg/kg IV

Day -4: Fludarabine 30 mg/m2 IV

Day -3: Fludarabine 30 mg/m2 IV

Day -2: Fludarabine 30 mg/m2 IV

Day -1: Total body irradiation (TBI) 200 centigray (cGy)

Day 0: Haploidentical bone marrow stem cell infusion

Day +3: Cyclophosphamide 50 mg/kg IV

Day +4: Cyclophosphamide 50 mg/kg IV

Day +5: Sirolimus (through day +365); mycophenolate mofetil (MMF) 15 mg/kg/dose three times per day (TID) (through day +35)

ELIGIBILITY:
Inclusion Criteria:

* Must weigh >25 kg at the time of study entry.
* Must have undergone puberty at the time of study entry to allow pre-transplant fertility preservation to occur, if desired. Puberty will be defined as Tanner III or more in male patients (typically age ≥ 13 years) and menarche in female patients.
* Have severe sickle cell disease (SCD) defined as 1 or more of the following:

  1. Clinically significant neurologic event (stroke) or any neurological deficit lasting > 24 hours;
  2. History of ≥2 episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea);
  3. History of ≥3 severe pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea);
  4. Administration of regular red blood cell (RBC) transfusion therapy, defined as receiving ≥8 transfusions per year for ≥1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome);
  5. An echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity ≥2.7 m/sec in adult patients.
* Have adequate physical function as measured by:

  1. Lansky or Karnofsky performance score ≥60
  2. Cardiac function: left ventricular ejection fraction (LVEF) >40% or LV shortening fraction > 26% by cardiac echocardiogram or by multigated acquisition (MUGA) scan.
  3. Pulmonary function: pulse oximetry with a baseline O2 saturation of ≥90% and DLCO >40% (corrected for hemoglobin)
  4. Renal function: serum creatinine ≤1.5 x the upper limit of normal for age as per local laboratory and 24 hour urine creatinine clearance >70 mL/min/1.73 m2 or glomerular filtration rate (GFR) >70 mL/min/1.73 m2 by radionuclide GFR.
  5. Hepatic function: serum conjugated (direct) bilirubin <2x upper limit of normal for age as per local laboratory and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5x upper limit of normal as per local laboratory. Patients with hyperbilirubinemia as a consequence of hyperhemolysis or who experience a sudden, profound change in the serum hemoglobin after a RBC transfusion are not excluded.
  6. In patients who have received chronic transfusion therapy for ≥1 year and who have clinical evidence of iron overload by serum ferritin or MRI, evaluation by liver biopsy is required. Histological examination of the liver must document the absence of cirrhosis, bridging fibrosis and active hepatitis. The absence of bridging fibrosis will be determined using the histological grading and staging scale as described by Ishak and colleagues (1995).
* Must be HLA typed at high resolution using DNA based typing at HLA-A, -B, -C and DRB1 and have an available related haploidentical bone marrow donor with 2, 3, or 4 (out of 8) HLA-mismatches. A unidirectional mismatch in either the graft versus host or host versus graft direction is considered a mismatch.

Exclusion Criteria:

* Availability of an 8 of 8 (HLA-A, B, C and DRB1) human leukocyte antigen (HLA) matched sibling or matched unrelated donor
* Presence of donor directed HLA antibodies.
* Severe pulmonary disease (despite above oxygen saturation and DLCO) including severe and uncontrolled asthma (per 2007 NHLBI Guidelines for the Diagnosis and Treatment of Asthma Expert Panel Report 3; http://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines/full-report), chronic obstructive pulmonary disease, and/or pulmonary hypertension (PH). A diagnosis of pulmonary hypertension (PH) will be made by finding of mean pulmonary artery pressure (mPAP) <25 mm Hg on right heart catheterization. In patients unable and/or unwilling to undergo cardiac catheterization, patients will be excluded with the following constellation of findings based upon presumptive diagnosis of PH (PPV of 62%): TRJ velocity >2.5 m/sec AND either N-terminal pro-brain natriuretic peptide (NT-pro-BNP) ≥160 pg/ml OR 6-minute walk distance <333 m.
* Uncontrolled bacterial, viral or fungal infection in the 6 week before enrollment
* Seropositivity for human immunodeficiency virus (HIV)
* Previous hematopoietic cell transplantation (HCT)
* Participation in a clinical trial in which the patient received an investigational drug or device or the off-label use of a drug or device within 3 months of enrollment
* Demonstrated lack of compliance with prior medical care
* Unwilling to use approved contraception for at least 6 months following transplant
* Pregnant or breastfeeding females
* Allergy to any component of mesenchymal stromal cell (MSC) suspension (such as human albumin) and/or allergy to any drugs used in HCT conditioning regimen.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of EPIC2016-MSC003 based upon dose limiting toxicities (DLTs) | 30 days after last MSC infusion
  DLTs will be defined as any grade ≥3 adverse reaction that is unexpected or considered attributable to the MSC infusion (attribution listed as at least probable). Because of the medical complexity of subjects on this trial and the lack of described DLTs to MSC infusion, all reported DLTs will be reviewed by the Data and Safety Monitoring Committee (DSMC).

SECONDARY OUTCOMES:
Primary graft rejection | 42 days after HCT
  Defined as the absence of donor cells assessed by peripheral blood chimerism assays on day 42.
Late graft rejection | One year after HCT
  Defined as the absence of donor hematopoietic cells in peripheral blood beyond day 42 in a patient who had initial evidence of hematopoietic recovery with > 20% donor cells.
Time to neutrophil engraftment | Up to one year after HCT
  Defined as the first of 3 measurements on different days when the patient has an absolute neutrophil count of 500/µL after conditioning.
Time to platelet engraftment | Up to one year after HCT
  Defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count > 50,000/µL AND did not receive a platelet transfusion in the previous 7 days.
Lineage specific donor chimerism | Up to one year after HCT
  Genomic deoxyribonucleic acid (DNA) extracted from peripheral blood will be analyzed for variable number of tandem repeats (VNTR) to detect donor engraftment in myeloid and lymphoid fractions.
Immune reconstitution | Up to one year after HCT
  Immune reconstitution will be assessed post-transplant by standard clinical testing and research testing.
Acute GVHD | One year after HCT
  Incidence of grade II-IV and III-IV acute GVHD
Chronic GVHD | One year after HCT
  Incidence and severity of chronic GVHD
Transplant-related mortality (TRM) | One year after HCT
  Defined as any death occurring in continuous complete remission
Event-free survival (EFS) | One year after HCT
  Defined as survival with stable donor erythropoiesis and no new clinical evidence SCD. Primary or late graft rejection with disease recurrence or death will count as events for this endpoint.
Overall survival (OS) | One year after HCT
  Defined as survival with or without SCD after HCT

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stenger, MD, Principal Investigator — Emory University; Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: No